CLINICAL TRIAL: NCT01975831
Title: A Phase 1 Study to Evaluate the Safety and Tolerability of Anti-PD-L1, MEDI4736, in Combination With Tremelimumab in Subjects With Advanced Solid Tumors
Brief Title: A Phase 1 Study to Evaluate MEDI4736 in Combination With Tremelimumab
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ludwig Institute for Cancer Research (Other)
Collaborators: MedImmune LLC (Industry); Cancer Research Institute, New York City (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LUD2013-003
Record Dates: First submitted 2013-10-29; First posted 2013-11-05 (Estimated); Results first posted 2020-06-22 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Breast Cancer; Ovarian Cancer; Colorectal Cancer; Cervical Cancer; Renal Cell Carcinoma
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms; Colorectal Neoplasms; Uterine Cervical Neoplasms; Carcinoma, Renal Cell | interventions — durvalumab; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Escalation: 0.3 mg/kg Durva + 3 mg/kg Treme (Experimental): Subjects received durvalumab (0.3 mg/kg every 2 weeks [Q2W] for 13 cycles) and tremelimumab (3 mg/kg every 4 weeks [Q4W] for 6 cycles, then every 12 weeks [Q12W]). Optional extended treatment comprised durvalumab monotherapy administered at the recommended fixed dose of 1500 mg Q4W.
  Interventions: Drug: Durvalumab; Drug: Tremelimumab
- Escalation: 1 mg/kg Durva + 3 mg/kg Treme (Experimental): Subjects received durvalumab (1 mg/kg Q2W for 13 cycles) and tremelimumab (3 mg/kg Q4W for 6 cycles, then Q12W). Optional extended treatment comprised durvalumab monotherapy administered at the recommended fixed dose of 1500 mg Q4W.
  Interventions: Drug: Durvalumab; Drug: Tremelimumab
- Escalation: 3 mg/kg Durva + 3 mg/kg Treme (Experimental): Subjects received durvalumab (3 mg/kg Q2W for 13 cycles) and tremelimumab (3 mg/kg Q4W for 6 cycles, then Q12W). Optional extended treatment comprised durvalumab monotherapy administered at the recommended fixed dose of 1500 mg Q4W.
  Interventions: Drug: Durvalumab; Drug: Tremelimumab
- Escalation: 3 mg/kg Durva + 1 mg/kg Treme (Experimental): Subjects received durvalumab (3 mg/kg Q2W for 12 or 13 cycles) and tremelimumab (1 mg/kg Q4W for 6 cycles, then Q12W or Q4W for 4 cycles). Optional extended treatment comprised durvalumab monotherapy administered at the recommended fixed dose of 1500 mg Q4W.
  Interventions: Drug: Durvalumab; Drug: Tremelimumab
- Expansion: Ovarian Cancer (Experimental): Subjects received durvalumab (10 mg/kg Q2W for 13 cycles or 1500 mg Q4W for 12 cycles) and tremelimumab (1 mg/kg or 75 mg Q4W for 4 cycles). Optional extended treatment comprised durvalumab monotherapy administered at the recommended fixed dose of 1500 mg Q4W.
  Interventions: Drug: Durvalumab; Drug: Tremelimumab
- Expansion: Colorectal Cancer (Experimental): Subjects received durvalumab (10 mg/kg Q2W for 13 cycles or 1500 mg Q4W for 12 cycles) and tremelimumab (1 mg/kg or 75 mg Q4W for 4 cycles). Optional extended treatment comprised durvalumab monotherapy administered at the recommended fixed dose of 1500 mg Q4W.
  Interventions: Drug: Durvalumab; Drug: Tremelimumab
- Expansion: Non-triple Negative Breast Cancer (Experimental): Subjects received durvalumab (10 mg/kg Q2W for 13 cycles or 1500 mg Q4W for 12 cycles) and tremelimumab (1 mg/kg or 75 mg Q4W for 4 cycles). Optional extended treatment comprised durvalumab monotherapy administered at the recommended fixed dose of 1500 mg Q4W.
  Interventions: Drug: Durvalumab; Drug: Tremelimumab
- Expansion: Renal Cell Carcinoma (Experimental): Subjects received durvalumab (10 mg/kg Q2W for 13 cycles or 1500 mg Q4W for 12 cycles) and tremelimumab (1 mg/kg or 75 mg Q4W for 4 cycles). Optional extended treatment comprised durvalumab monotherapy administered at the recommended fixed dose of 1500 mg Q4W.
  Interventions: Drug: Durvalumab; Drug: Tremelimumab
- Expansion: Cervical Cancer (Experimental): Subjects received durvalumab (10 mg/kg Q2W for 13 cycles or 1500 mg Q4W for 12 cycles) and tremelimumab (1 mg/kg or 75 mg Q4W for 4 cycles). Optional extended treatment comprised durvalumab monotherapy administered at the recommended fixed dose of 1500 mg Q4W.
  Interventions: Drug: Durvalumab; Drug: Tremelimumab

INTERVENTIONS:
Drug: Durvalumab — Durvalumab was administered as an intravenous (IV) infusion over 60 (± 5) minutes.
  Other Names: MEDI4736; Durva
Drug: Tremelimumab — Tremelimumab was administered as an intravenous (IV) infusion over 60 (± 5) minutes.
  Other Names: Treme

SUMMARY:
This was a Phase 1, open-label, nonrandomized, multicenter study of durvalumab and tremelimumab in subjects with advanced cancers who were not eligible for, declined, or failed standard treatment. The primary study objective was to determine the maximum tolerated dose (MTD) and safety profile of the durvalumab and tremelimumab combination. Secondary objectives were to evaluate the pharmacokinetics (PK) and immunogenicity of durvalumab and tremelimumab, and the antitumor activity (tumor response, progression-free survival [PFS], and overall survival [OS]) of the durvalumab and tremelimumab combination. (Note: Collection of PK and immunogenicity samples was removed by amendment; analysis was not done.) Exploratory objectives were to evaluate the biological activity of the durvalumab and tremelimumab combination.

DETAILED DESCRIPTION:
The study comprised a 3 + 3 dose escalation phase in which 3 to 6 subjects were enrolled into sequential cohorts until determination of the MTD, followed by an expansion phase in 5 tumor type-specific cohorts (i.e., ovarian cancer, colorectal cancer, non-triple negative breast cancer, renal cell carcinoma, and cervical cancer). Each expansion cohort was to include 15 subjects treated with the identified MTD or maximum dose tested in the dose-escalation phase.

Subjects received durvalumab and tremelimumab over 12 to 13 four-week cycles during the Core Study, with continuous monitoring for safety, clinical efficacy, and biological activity, followed by optional treatment extension with durvalumab for subjects maintaining at least stable disease if agreed upon by the Investigator and Sponsor. After study treatment completion, study assessments were continued for up to 90 days after the last administration of study treatment or until start of alternate therapy, with long-term follow up after study completion for clinical outcomes at least every 6 months for up to 3 years following initiation of treatment.

Study treatment in the Core Study continued for up to 12 months or until confirmed progressive disease (PD), initiation of alternative cancer therapy, observation of unacceptable toxicity, or any other criteria for treatment discontinuation.

Optional treatment extension beyond the Core Study was permitted for subjects who completed the Core Study with a tumor response of stable disease or better and upon agreement by the Sponsor and Investigator. Extended treatment comprised durvalumab monotherapy administered at the recommended fixed dose of 1500 mg administered every 4 weeks (Q4W).

ELIGIBILITY:
Inclusion Criteria

1. Histologically- or cytologically-confirmed ovarian cancer, colorectal cancer, non-triple negative breast cancer, renal cell carcinoma and cervical cancer, with at least one lesion measurable by the immune-related Response Criteria (irRC) not previously irradiated. NOTE: Per Amendment 5, the disease states of non-small cell lung cancer and head and neck cancer were removed from the study and were replaced by non-triple negative breast cancer.
2. Failed to respond to or relapsed following standard treatment or declined or was not eligible for standard treatment.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2.
4. Anticipated lifespan greater than 6 months.
5. At the time of Day 1 of the study, subjects with brain metastases must have been asymptomatic for at least 4 weeks and:

   * at least 8 weeks without tumor progression after any whole brain radiotherapy;
   * at least 4 weeks since craniotomy and resection or stereotactic radiosurgery;
   * at least 3 weeks without new brain metastases as evidenced by magnetic resonance imaging (MRI)/computed tomography (CT).
6. Adequate organ and marrow function, as defined below:

   * hemoglobin ≥ 9 g/dL
   * absolute neutrophil count ≥ 1500/mm^3
   * platelet count ≥ 100,000/mm^3
   * total bilirubin within normal ranges unless associated with hepatobiliary metastases or Gilbert syndrome, then total bilirubin ≤ 2 × the upper limit of normal (ULN)
   * alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN unless associated with hepatic metastases, then ALT and AST ≤ 5 × ULN
   * creatinine ≤ 2.0 mg/dL
7. Have been informed of other treatment options.
8. Age ≥ 18 years.
9. Able and willing to give valid written informed consent.
10. Able and willing to give valid written consent for archival tumor samples.
11. Able and willing to give valid written consent for biopsy samples (subjects with biopsiable tumors, and if clinically appropriate, in the expansion phase only).

Exclusion Criteria

1. Prior exposure to tremelimumab or durvalumab or other anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4), anti-programmed cell death-1 (PD-1), anti-programmed cell death ligand-1 (PD-L1) antibodies.
2. History of severe allergic reactions to any unknown allergens or any components of the study drugs.
3. Active or prior autoimmune disease except for autoimmune thyroiditis or vitiligo.
4. Any prior Grade ≥ 3 immune-related adverse event (irAE) or any prior corticosteroid-refractory irAE.
5. Known active or chronic viral hepatitis or history of any type of hepatitis within the last 6 months.
6. History of sarcoidosis syndrome.
7. Active or history of inflammatory bowel disease (colitis, Crohn's), diverticulitis, irritable bowel disease, celiac disease, or other serious, chronic, gastrointestinal conditions associated with diarrhea. Active or history of systemic lupus erythematosus or Wegener's granulomatosis.
8. Metastatic disease to the central nervous system for which other therapeutic options, including radiotherapy, may have been available.
9. Known immunodeficiency or active human immunodeficiency virus (HIV).
10. Other active serious illnesses (e.g., serious infections requiring antibiotics).
11. If a subject previously received investigational treatment, the last dose of investigational treatment was administered within 4 weeks of Day 1 of the study or AE(s) attributable to investigational treatment had not resolved to Grade 1 or better.
12. Major surgical procedure (as defined by the Investigator) within 30 days prior to Day 1 or still recovering from prior surgery.
13. Mental impairment that may have compromised the ability to give informed consent and comply with the requirements of the study.
14. Lack of availability for immunological and clinical follow-up assessments.
15. Women who were breast feeding or pregnant as evidenced by positive serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]).
16. Female subjects of childbearing potential who were sexually active with a non-sterilized male partner must have used at least one highly effective method of contraception from the time of screening and must have agreed to continue using such precautions for 90 days after the last dose of durvalumab or for 6 months after the final dose of durvalumab + tremelimumab (whichever was longer). Non-sterilized male partners of a female subject must have used male condoms plus spermicide throughout this period. Cessation of birth control after this point should have been discussed with a responsible physician. Not engaging in sexual activity for the total duration of the trial and the drug washout period was an acceptable practice; however, periodic abstinence, the rhythm method, and the withdrawal method were not acceptable methods of birth control.

    Female subjects should have also refrained from breastfeeding throughout the period described above.

    Females of childbearing potential were defined as those who were not surgically sterile (i.e., bilateral tubal ligation, bilateral oophorectomy, or complete hysterectomy) or post-menopausal.

    Females were considered post-menopausal if they had been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements applied:
    * Females <50 years of age were considered post-menopausal if they had been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they had luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
    * Females ≥ 50 years of age were considered post-menopausal if they had been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).

    Non-sterilized male subjects who were sexually active with a female partner of childbearing potential must have used male condoms plus spermicide from screening through 90 days after the last dose of durvalumab or through 6 months after receipt of the final dose of durvalumab + tremelimumab (whichever was longer). Female partners (of childbearing potential) of a male subject must have used a highly effective method of contraception throughout this period. Cessation of birth control after this point should have been discussed with a responsible physician. Not engaging in sexual activity for the total duration of the trial and the drug washout period was an acceptable practice; however, periodic abstinence, the rhythm method, and the withdrawal method were not acceptable methods of contraception.

    Male subjects should have refrained from sperm donation throughout the period described above.

    A highly effective method of contraception was defined as one that resulted in a low failure rate (i.e. less than 1% per year) when used consistently and correctly. Note that some contraception methods were not considered highly effective (e.g., male or female condom with or without spermicide; female cap, diaphragm, or sponge with or without spermicide; non-copper containing intrauterine device; progestogen-only oral hormonal contraceptive pills where inhibition of ovulation is not the primary mode of action [excluding Cerazette/desogestrel which was considered highly effective]; and triphasic combined oral contraceptive pills).
17. Any condition that, in the clinical judgment of the treating physician, was likely to prevent the subject from complying with any aspect of the protocol or that may have put the subject at unacceptable risk.
18. Subjects must not have donated blood while on study and for at least 90 days following the last durvalumab treatment or 6 months after the last tremelimumab treatment, whichever was longer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2013-12-19 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2021-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jedd D Wolchok, MD, PhD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (6):
- United States (6):
  - Yale Cancer Center, New Haven, Connecticut
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Mary Crowley Cancer Research Center, Dallas, Texas
  - University of Virginia Division of Hematology and Oncology, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wolchok JD, Hoos A, O'Day S, Weber JS, Hamid O, Lebbe C, Maio M, Binder M, Bohnsack O, Nichol G, Humphrey R, Hodi FS. Guidelines for the evaluation of immune therapy activity in solid tumors: immune-related response criteria. Clin Cancer Res. 2009 Dec 1;15(23):7412-20. doi: 10.1158/1078-0432.CCR-09-1624. Epub 2009 Nov 24. PMID 19934295
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774

RESULTS

PARTICIPANT FLOW:
Groups:
- Escalation: 0.3 mg/kg Durva + 3 mg/kg Treme: Subjects received durvalumab (0.3 mg/kg every 2 weeks [Q2W] for 13 cycles) and tremelimumab (3 mg/kg every 4 weeks [Q4W] for 6 cycles, then every 12 weeks [Q12W]). Optional extended treatment comprised durvalumab monotherapy administered at the recommended fixed dose of 1500 mg Q4W.
  Durvalumab and tremelimumab were administered as intravenous (IV) infusions over 60 (± 5) minutes, with durvalumab infusions started at least 60 minutes after the end of the tremelimumab infusion on dual dosing days.
- Escalation: 1 mg/kg Durva + 3 mg/kg Treme: Subjects received durvalumab (1 mg/kg Q2W for 13 cycles) and tremelimumab (3 mg/kg Q4W for 6 cycles, then Q12W). Optional extended treatment comprised durvalumab monotherapy administered at the recommended fixed dose of 1500 mg Q4W.
  Durvalumab and tremelimumab were administered as IV infusions over 60 (± 5) minutes, with durvalumab infusions started at least 60 minutes after the end of the tremelimumab infusion on dual dosing days.
- Escalation: 3 mg/kg Durva + 3 mg/kg Treme: Subjects received durvalumab (3 mg/kg Q2W for 13 cycles) and tremelimumab (3 mg/kg Q4W for 6 cycles, then Q12W). Optional extended treatment comprised durvalumab monotherapy administered at the recommended fixed dose of 1500 mg Q4W.
  Durvalumab and tremelimumab were administered as IV infusions over 60 (± 5) minutes, with durvalumab infusions started at least 60 minutes after the end of the tremelimumab infusion on dual dosing days.
- Escalation: 3 mg/kg Durva + 1 mg/kg Treme: Subjects received durvalumab (3 mg/kg Q2W for 12 or 13 cycles) and tremelimumab (1 mg/kg Q4W for 6 cycles, then Q12W or Q4W for 4 cycles). Optional extended treatment comprised durvalumab monotherapy administered at the recommended fixed dose of 1500 mg Q4W.
  Durvalumab and tremelimumab were administered as IV infusions over 60 (± 5) minutes, with durvalumab infusions started at least 60 minutes after the end of the tremelimumab infusion on dual dosing days.
- Expansion: Ovarian Cancer; Expansion: Colorectal Cancer; Expansion: Non-triple Negative Breast Cancer; Expansion: Renal Cell Carcinoma; Expansion: Cervical Cancer: Subjects received durvalumab (10 mg/kg Q2W for 13 cycles or 1500 mg Q4W for 12 cycles) and tremelimumab (1 mg/kg or 75 mg Q4W for 4 cycles). Optional extended treatment comprised durvalumab monotherapy administered at the recommended fixed dose of 1500 mg Q4W.
  Durvalumab and tremelimumab were administered as IV infusions over 60 (± 5) minutes, with durvalumab infusions started at least 60 minutes after the end of the tremelimumab infusion on dual dosing days.
Period: Overall Study
Arm/Group | Escalation: 0.3 mg/kg Durva + 3 mg/kg Treme | Escalation: 1 mg/kg Durva + 3 mg/kg Treme | Escalation: 3 mg/kg Durva + 3 mg/kg Treme | Escalation: 3 mg/kg Durva + 1 mg/kg Treme | Expansion: Ovarian Cancer | Expansion: Colorectal Cancer | Expansion: Non-triple Negative Breast Cancer | Expansion: Renal Cell Carcinoma | Expansion: Cervical Cancer
Started | 3 | 11 | 4 | 4 | 19 | 16 | 16 | 16 | 15
Completed | 0 | 2 | 0 | 0 | 1 | 2 | 0 | 1 | 3
Not Completed | 3 | 9 | 4 | 4 | 18 | 14 | 16 | 15 | 12
Not completed — Adverse Event | 1 | 2 | 2 | 0 | 1 | 1 | 3 | 4 | 1
Not completed — Death | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Progressive Disease | 1 | 3 | 2 | 4 | 13 | 9 | 10 | 8 | 10
Not completed — Withdrawal by Subject | 0 | 3 | 0 | 0 | 3 | 1 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Initiation of Subsequent Therapy | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Not completed — Entered Hospice | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Unable to Treat Within Protocol Windows | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The population comprises all subjects who received any dose of study treatment.
Groups:
- Escalation: 0.3 mg/kg Durva + 3 mg/kg Treme: Subjects received durvalumab (0.3 mg/kg Q2W for 13 cycles) and tremelimumab (3 mg/kg Q4W for 6 cycles, then Q12W). Optional extended treatment comprised durvalumab monotherapy administered at the recommended fixed dose of 1500 mg Q4W.
  Durvalumab and tremelimumab were administered as IV infusions over 60 (± 5) minutes, with durvalumab infusions started at least 60 minutes after the end of the tremelimumab infusion on dual dosing days.
- Total: Total of all reporting groups
Arm/Group | Escalation: 0.3 mg/kg Durva + 3 mg/kg Treme | Escalation: 1 mg/kg Durva + 3 mg/kg Treme | Escalation: 3 mg/kg Durva + 3 mg/kg Treme | Escalation: 3 mg/kg Durva + 1 mg/kg Treme | Expansion: Ovarian Cancer | Expansion: Colorectal Cancer | Expansion: Non-triple Negative Breast Cancer | Expansion: Renal Cell Carcinoma | Expansion: Cervical Cancer | Total
Number analyzed (Participants) | 3 | 11 | 4 | 4 | 19 | 16 | 16 | 16 | 15 | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (7.51) | 54.9 (11.93) | 50.3 (10.21) | 52.8 (11.35) | 59.7 (10.91) | 49.7 (9.79) | 55.4 (14.31) | 59.7 (9.71) | 53.0 (11.46) | 55.5 (11.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 3 | 3 | 19 | 9 | 16 | 2 | 15 | 76
  Male | 0 | 5 | 1 | 1 | 0 | 7 | 0 | 14 | 0 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 5
  Not Hispanic or Latino | 3 | 10 | 3 | 4 | 17 | 14 | 14 | 16 | 12 | 93
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 1 | 3 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Black or African American | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 2 | 5
  White | 3 | 10 | 2 | 4 | 16 | 12 | 12 | 15 | 9 | 83
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 0 | 0 | 2 | 2 | 0 | 1 | 7
Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) [Count of Participants; unit: Participants] — PS 0 = Fully active, able to carry on all pre-disease performance without restriction; PS 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; PS 2 = Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours; PS 3 = Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours; PS 4 = Completely disabled; cannot carry on any selfcare; totally confined to bed or chair; PS 5 = Dead
  Participants
    ECOG PS 0 | 2 | 2 | 2 | 1 | 7 | 9 | 6 | 14 | 9 | 52
    ECOG PS 1 | 1 | 9 | 2 | 2 | 11 | 7 | 10 | 2 | 6 | 50
    ECOG PS 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Treatment-emergent Adverse Events (TEAEs)
Description: Toxicity was graded in accordance with the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.03. Adverse events (AEs) were reported based on clinical laboratory tests, vital sign and weight measurements, physical examinations, performance status evaluations, electrocardiograms, magnetic resonance imaging, and any other medically indicated assessments, including subject interviews, from the time informed consent is signed through 90 days after the last dose of study treatment. AEs were considered to be treatment emergent (TEAE) if they occurred or worsened in severity after the first dose of study treatment.
Time Frame: Up to 36 months
Population: The population comprises all subjects who received any dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Escalation: 0.3 mg/kg Durva + 3 mg/kg Treme | Escalation: 1 mg/kg Durva + 3 mg/kg Treme | Escalation: 3 mg/kg Durva + 3 mg/kg Treme | Escalation: 3 mg/kg Durva + 1 mg/kg Treme | Expansion: Ovarian Cancer | Expansion: Colorectal Cancer | Expansion: Non-triple Negative Breast Cancer | Expansion: Renal Cell Carcinoma | Expansion: Cervical Cancer
Number analyzed (Participants) | 3 | 11 | 4 | 4 | 19 | 16 | 16 | 16 | 15
Participants
  Any TEAE | 3 | 11 | 4 | 4 | 19 | 16 | 16 | 16 | 15
  Serious TEAE | 2 | 5 | 4 | 1 | 9 | 8 | 8 | 6 | 8
  TEAE leading to treatment discontinuation | 1 | 4 | 2 | 0 | 4 | 1 | 4 | 4 | 2

2. Secondary Outcome: Number of Subjects With Best Overall Immune-related Tumor Response
Description: Immune-related tumor response was evaluated by computed tomography at Baseline and every 4 to 8 or 12 weeks on study. Tumor response was designated according to the immune-related Response Criteria (irRC) (Wolchok et al 2009) into the following categories: immune-related complete response (irCR) requires disappearance of all lesions in two consecutive observations not less than 4 weeks apart; immune-related partial response (irPR) requires ≥ 50% decrease in tumor burden compared with baseline in two observations at least 4 weeks apart; immune-related stable disease (irSD) is assigned when neither a 50% decrease from baseline tumor burden nor a 25% increase in tumor burden from nadir can be established; immune-related progressive disease (irPD) requires a ≥ 25% increase from nadir in tumor burden at any single time point in two consecutive observations at least 4 weeks apart.
Time Frame: Up to 24 months
Population: The population comprises all subjects who received at least one dose of the durvalumab/tremelimumab combination and had the baseline and at least one post-baseline assessment of any efficacy endpoint (clinical or radiological) or a report of death.
Measure: Count of Participants; unit: Participants
Arm/Group | Escalation: 0.3 mg/kg Durva + 3 mg/kg Treme | Escalation: 1 mg/kg Durva + 3 mg/kg Treme | Escalation: 3 mg/kg Durva + 3 mg/kg Treme | Escalation: 3 mg/kg Durva + 1 mg/kg Treme | Expansion: Ovarian Cancer | Expansion: Colorectal Cancer | Expansion: Non-triple Negative Breast Cancer | Expansion: Renal Cell Carcinoma | Expansion: Cervical Cancer
Number analyzed (Participants) | 3 | 10 | 3 | 4 | 18 | 15 | 16 | 15 | 15
Participants
  irCR | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  irPR | 0 | 2 | 0 | 0 | 1 | 1 | 1 | 2 | 3
  irSD | 2 | 3 | 1 | 0 | 7 | 1 | 2 | 11 | 3
  irPD | 1 | 5 | 2 | 4 | 10 | 12 | 12 | 2 | 7
  Not evaluable | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1

3. Secondary Outcome: Number of Subjects With Best Overall Tumor Response by Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Description: Tumor response was evaluated using computed tomography and categorized according to RECIST (version 1.1) at Baseline and every 4 to 8 or 12 weeks on study. Per RECIST 1.1 (Eisenhauer et al 2009), target lesions are categorized as follows: Complete Response (CR): Disappearance of all target lesions; Partial Response (PR): ≥ 30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD): ≥ 20% increase in the sum of the longest diameter of target lesions; Stable Disease (SD): small changes that do not meet above criteria.
Time Frame: Up to 24 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Escalation: 0.3 mg/kg Durva + 3 mg/kg Treme | Escalation: 1 mg/kg Durva + 3 mg/kg Treme | Escalation: 3 mg/kg Durva + 3 mg/kg Treme | Escalation: 3 mg/kg Durva + 1 mg/kg Treme | Expansion: Ovarian Cancer | Expansion: Colorectal Cancer | Expansion: Non-triple Negative Breast Cancer | Expansion: Renal Cell Carcinoma | Expansion: Cervical Cancer
Number analyzed (Participants) | 3 | 10 | 3 | 4 | 18 | 15 | 16 | 15 | 15
Participants
  CR | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  PR | 0 | 2 | 0 | 0 | 1 | 1 | 1 | 3 | 3
  SD | 2 | 3 | 1 | 0 | 6 | 1 | 4 | 7 | 3
  PD | 1 | 5 | 2 | 4 | 11 | 12 | 11 | 5 | 8

4. Secondary Outcome: Median Progression-free Survival Per irRC Based on Kaplan-Meier Product Limit Estimates
Description: PFS was measured from the date of the first dose of study treatment to the date of the first confirmed progression (including clinical progression) or the date of death if a subject died before progression. Per irRC, irPD requires a ≥ 25% increase from nadir in tumor burden at any single time point in two consecutive observations at least 4 weeks apart (Wolchok et al 2009). Subjects who did not experience a PFS event (progression or death) were censored at the date of the last tumor assessment. Subjects with no relevant tumor response assessment were censored at the start date of study treatment.
Time Frame: Up to 36 months
Population: as for outcome 2
Measure: Median (Full Range); unit: days
Arm/Group | Escalation: 0.3 mg/kg Durva + 3 mg/kg Treme | Escalation: 1 mg/kg Durva + 3 mg/kg Treme | Escalation: 3 mg/kg Durva + 3 mg/kg Treme | Escalation: 3 mg/kg Durva + 1 mg/kg Treme | Expansion: Ovarian Cancer | Expansion: Colorectal Cancer | Expansion: Non-triple Negative Breast Cancer | Expansion: Renal Cell Carcinoma | Expansion: Cervical Cancer
Number analyzed (Participants) | 3 | 10 | 3 | 4 | 18 | 15 | 16 | 15 | 15
days | 82 [48 to 82] | 76 [34 to 1007] | 51 [49 to 401] | 42 [40 to 52] | 54 [12 to 618] | 57 [32 to 559] | 57 [27 to 223] | 326 [54 to 611] | 79 [32 to 617]

5. Secondary Outcome: Median Progression-free Survival Per RECIST 1.1 Based on Kaplan-Meier Product Limit Estimates
Description: PFS was measured from the date of the first dose of study treatment to the date of the first confirmed progression (including clinical progression) or the date of death if a subject died before progression. Per RECIST 1.1, PD requires a ≥ 20% increase in the sum of the longest diameter of target lesions (Eisenhauer et al 2009). Subjects who did not experience a PFS event (progression or death) were censored at the date of the last tumor assessment. Subjects with no relevant tumor response assessment were censored at the start date of study treatment.
Time Frame: Up to 36 months
Population: as for outcome 2
Measure: Median (Full Range); unit: days
Arm/Group | Escalation: 0.3 mg/kg Durva + 3 mg/kg Treme | Escalation: 1 mg/kg Durva + 3 mg/kg Treme | Escalation: 3 mg/kg Durva + 3 mg/kg Treme | Escalation: 3 mg/kg Durva + 1 mg/kg Treme | Expansion: Ovarian Cancer | Expansion: Colorectal Cancer | Expansion: Non-triple Negative Breast Cancer | Expansion: Renal Cell Carcinoma | Expansion: Cervical Cancer
Number analyzed (Participants) | 3 | 10 | 3 | 4 | 18 | 15 | 16 | 15 | 15
days | 82 [48 to 251] | 76 [34 to 1007] | 51 [49 to 401] | 42 [40 to 52] | 54 [12 to 618] | 57 [32 to 559] | 56 [27 to 223] | 279 [50 to 555] | 58 [27 to 617]

6. Secondary Outcome: Median Overall Survival (OS) Based on Kaplan-Meier Product Limit Estimates
Description: All subjects were monitored for survival follow-up at least every 6 months after study completion for up to 3 years after initiation of treatment. Subjects who continued into the Extension part of the study may have been followed for longer than 3 years if they were still receiving treatment. OS was measured from the date of the first dose of study treatment until the recorded date of death. Subjects without a recorded outcome of death were censored at the date of last contact.
Time Frame: Up to 48 months
Population: as for outcome 2
Measure: Median (Full Range); unit: days
Arm/Group | Escalation: 0.3 mg/kg Durva + 3 mg/kg Treme | Escalation: 1 mg/kg Durva + 3 mg/kg Treme | Escalation: 3 mg/kg Durva + 3 mg/kg Treme | Escalation: 3 mg/kg Durva + 1 mg/kg Treme | Expansion: Ovarian Cancer | Expansion: Colorectal Cancer | Expansion: Non-triple Negative Breast Cancer | Expansion: Renal Cell Carcinoma | Expansion: Cervical Cancer
Number analyzed (Participants) | 3 | 10 | 3 | 4 | 18 | 15 | 16 | 15 | 15
days | 321 [48 to 482] | 592 [44 to 1380] | 664 [76 to 1000] | 223 [120 to 873] | 460 [12 to 652] | 267 [56 to 559] | 267 [35 to 589] | 462 [312 to 611] | 583 [32 to 617]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were documented from informed consent through 90 days after the last study drug dose (regardless of causality to study drug), i.e., during the treatment period, which was up to 15 months for those participating in the Core Study and up to 36 months for those continuing in the Extension. All-cause mortality was collected as a part of survival follow-up for up to 3 years after initiation of treatment, or longer (i.e., up to 48 months) for patients continuing in the Extension.
Description: AE documentation included onset/resolution dates, severity using the NCI CTCAE (version 4.03), seriousness, relationship to study drug, study drug action taken, treatment, and outcome. In summaries, preferred terms were counted only once per subject at the maximum reported grade.
Arm/Group | Escalation: 0.3 mg/kg Durva + 3 mg/kg Treme | Escalation: 1 mg/kg Durva + 3 mg/kg Treme | Escalation: 3 mg/kg Durva + 3 mg/kg Treme | Escalation: 3 mg/kg Durva + 1 mg/kg Treme | Expansion: Ovarian Cancer | Expansion: Colorectal Cancer | Expansion: Non-triple Negative Breast Cancer | Expansion: Renal Cell Carcinoma | Expansion: Cervical Cancer
All-Cause Mortality (participants affected / at risk) | 3/3 | 6/11 | 4/4 | 3/4 | 10/19 | 11/16 | 9/16 | 4/16 | 7/15
Serious Adverse Events (participants affected / at risk) | 2/3 | 5/11 | 4/4 | 1/4 | 9/19 | 8/16 | 8/16 | 6/16 | 8/15
Other Adverse Events (participants affected / at risk) | 3/3 | 11/11 | 4/4 | 4/4 | 19/19 | 16/16 | 16/16 | 16/16 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Escalation: 0.3 mg/kg Durva + 3 mg/kg Treme (N=3) | Escalation: 1 mg/kg Durva + 3 mg/kg Treme (N=11) | Escalation: 3 mg/kg Durva + 3 mg/kg Treme (N=4) | Escalation: 3 mg/kg Durva + 1 mg/kg Treme (N=4) | Expansion: Ovarian Cancer (N=19) | Expansion: Colorectal Cancer (N=16) | Expansion: Non-triple Negative Breast Cancer (N=16) | Expansion: Renal Cell Carcinoma (N=16) | Expansion: Cervical Cancer (N=15)
Nausea (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 1 | 3 | 1 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 3
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Duodenal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3 | 0 | 0 | 3 | 3 | 0 | 0 | 1
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Asthenia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Multi-organ failure (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Cardiac disorder (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vaginal fistula (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Kidney infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vulvitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Face oedema (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypothalamo-pituitary disorder (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Escalation: 0.3 mg/kg Durva + 3 mg/kg Treme (N=3) | Escalation: 1 mg/kg Durva + 3 mg/kg Treme (N=11) | Escalation: 3 mg/kg Durva + 3 mg/kg Treme (N=4) | Escalation: 3 mg/kg Durva + 1 mg/kg Treme (N=4) | Expansion: Ovarian Cancer (N=19) | Expansion: Colorectal Cancer (N=16) | Expansion: Non-triple Negative Breast Cancer (N=16) | Expansion: Renal Cell Carcinoma (N=16) | Expansion: Cervical Cancer (N=15)
Fatigue (General disorders) | 1 | 5 | 2 | 3 | 11 | 8 | 7 | 8 | 7
Nausea (Gastrointestinal disorders) | 0 | 3 | 1 | 1 | 3 | 3 | 6 | 5 | 3
Diarrhoea (Gastrointestinal disorders) | 1 | 8 | 0 | 2 | 8 | 4 | 7 | 1 | 3
Decreased appetite (Metabolism and nutrition disorders) | 1 | 5 | 1 | 0 | 4 | 5 | 4 | 5 | 5
Vomiting (Gastrointestinal disorders) | 0 | 5 | 2 | 0 | 7 | 6 | 4 | 2 | 4
Constipation (Gastrointestinal disorders) | 1 | 5 | 0 | 0 | 2 | 5 | 4 | 3 | 5
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 3 | 5 | 3 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2 | 2 | 1 | 4 | 3 | 2 | 3 | 3
Pyrexia (General disorders) | 0 | 1 | 1 | 0 | 2 | 2 | 1 | 2 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1 | 0 | 4 | 2 | 3 | 3 | 2
Oedema peripheral (General disorders) | 2 | 3 | 1 | 0 | 2 | 3 | 3 | 3 | 3
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 0 | 1 | 2 | 1 | 4 | 3 | 2
Anaemia (Blood and lymphatic system disorders) | 2 | 6 | 0 | 1 | 3 | 1 | 3 | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 0 | 3 | 2 | 3 | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 4 | 2 | 2 | 2 | 2
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 0 | 1 | 3 | 0 | 4 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 1 | 4 | 0 | 1 | 5 | 1
Weight decreased (Investigations) | 0 | 3 | 0 | 0 | 4 | 3 | 1 | 1 | 2
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 3 | 3 | 2 | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 2 | 3 | 3 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 2 | 0 | 0 | 2 | 3 | 1 | 2 | 2
Urinary tract infection (Infections and infestations) | 0 | 2 | 0 | 0 | 1 | 2 | 0 | 0 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 5 | 1 | 1 | 2 | 2 | 1 | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 0 | 3 | 2 | 2 | 0 | 2
Insomnia (Psychiatric disorders) | 0 | 1 | 1 | 1 | 4 | 3 | 1 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 2 | 0 | 1 | 1 | 0 | 2 | 2 | 2
Asthenia (General disorders) | 0 | 4 | 1 | 0 | 2 | 1 | 2 | 0 | 1
Chills (General disorders) | 1 | 2 | 1 | 1 | 1 | 1 | 1 | 2 | 2
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 0 | 3 | 3 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 2 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 2 | 2 | 1 | 1 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 3 | 1 | 0 | 1 | 1 | 0 | 1 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0 | 1 | 2 | 2 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 3 | 0 | 0 | 2 | 1 | 2 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1
Ascites (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 2 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 3 | 0 | 1 | 0 | 0
Malaise (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 3 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 1 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 1
Headache (Nervous system disorders) | 1 | 1 | 1 | 0 | 0 | 2 | 1 | 0 | 1
Hypotension (Vascular disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 3 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 2
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Device occlusion (General disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Early satiety (General disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Hypertension (Vascular disorders) | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Infusion site reaction (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 0
Vaginal fistula (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bladder spasm (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Mental status changes (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Swelling (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abscess oral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Akathisia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bacteriuria (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bilirubin conjugated increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood sodium decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Contrast media allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Euphoric mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypophysitis (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Irritability (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Livedo reticularis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Localised oedema (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lyme disease (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Monoplegia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neutrophil count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Onychomycosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pelvic discomfort (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Polydipsia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rectal tenesmus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Salivary gland calculus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sensory disturbance (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin striae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Speech disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Thirst (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tinea pedis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urine abnormality (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vaginal disorder (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paralysis (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Face oedema (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tenderness (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urine output decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Genital herpes (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mucosal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia staphylococcal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eye irritation (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Facial pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-08): https://cdn.clinicaltrials.gov/large-docs/31/NCT01975831/Prot_SAP_000.pdf